CLINICAL TRIAL: NCT00356850
Title: Ocular Pharmacokinetics After a Single Drop Instillation, in Each Eye of One of Three Different Concentrations of T1225 (0.5% - 1% - 1.5% Dihydrate) in 91 Healthy Volunteers
Brief Title: Ocular Pharmacokinetics After a Single Drop Instillation of T1225 0.5, 1, 1.5% in 91 Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT1225-PI2-03/02(F)
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-07

CONDITIONS: Eye Infections, Bacterial
MeSH Terms: conditions — Eye Infections, Bacterial | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To evaluate azithromycin tear concentrations after instillation of one drop of one of the three T1225 concentrations (0.5%, 1% and 1.5%) and to evaluate the ocular safety.

DETAILED DESCRIPTION:
The aim of the present study was to compare azithromycin tear ocular concentrations after a single instillation of three different T1225 concentrations in order to determine early azithromycin tear concentration and to assess the T1225 concentration, which allowed having the higher azithromycin tear concentration, 24 hours after a single instillation.

ELIGIBILITY:
Inclusion Criteria:

* Male/female aged from 18 to 45 years;
* Written informed consent;
* Healthy volunteers without any subjective ocular symptom;
* Corrected visual acuity >= 6/10;
* Registered in the national register of healthy volunteers

Exclusion Criteria:

* Ocular trauma, infection or inflammation within the last 3 months;
* Conjunctival hyperaemia (score >= 2);
* Folliculo-papillary conjunctivitis (score >= 2);
* Topical ocular treatment within the last month;
* Ocular surgery, including LASIK and PRK, within the last 12 months;
* Other ocular laser within the last 3 months;
* Zithromax® and Azadose® within the last 3 months;
* Medication during the study (except: paracetamol, contraceptives

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2002-05; Study Completion 2002-06

PRIMARY OUTCOMES:
Area Under the Curve from 0 to 24 hours (AUC0-24h)
Elimination half-life (t1/2)
Maximum Concentration (Cmax)
Concentration 24 hours after instillation (C24h)

SECONDARY OUTCOMES:
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Professor, Principal Investigator — Centre de Pharmacologie Clinique - Clermont-Ferrand (France)